CLINICAL TRIAL: NCT07266285
Title: A Phase 1 Trial of BTM-3566 in Advanced Solid Tumors
Brief Title: BTM-3566 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bantam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTM-3566-001-ST
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Phase 1; Dose escalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BTM-3566 (Experimental): Daily oral dosing (7 days on/7 days off)
  Interventions: Drug: BTM-3566

INTERVENTIONS:
Drug: BTM-3566 — BTM-3566

SUMMARY:
The goal of this clinical trial is to learn about what doses of BTM-356 are safe to use in adults with advanced cancers in solid tumors. It will also learn about how effective different doses of BTM-3566 are in treating cancer. The main questions it aims to answer are:

What adverse events and toxicities (harmful side effects) are associated with different doses of BTM-3566? What are the blood levels of BTM-3566 in your body at different timepoints? What effect does BTM-3566 have on reducing tumor size and/or preventing the worsening of cancer? All participants will receive BTM-3566 and none will receive placebo (a look-alike substance that contains no drug).

Participants will:

* Take BTM-3566 for 7 days, then take a 7 day break. This 2 week dosing schedule of 7 days on/7 days off will continue until your disease worsens or you cannot tolerate treatment.
* Visit the clinic approximately 7 times during screening and the first month of treatment. Visits will be reduced to approximately 2 visits per month after.
* Keep a diary of when (and how much) BTM-3566 you take, along with how much you weigh on each dosing day.

DETAILED DESCRIPTION:
This study is a phase 1, open label, dose escalation study using single participant cohorts followed by 3+3 design to evaluate multiple ascending doses of BTM-3566.

ELIGIBILITY:
Key Inclusion Criteria:

* Any advanced, unresectable and/or metastatic solid tumors except for primary brain cancer, breast cancer, prostate cancer, pancreatic cancer, pheochromocytoma, fibrolamellar carcinoma, adrenocortical carcinoma, or ocular or cutaneous melanoma.
* Must be refractory/relapsed after all standard therapies known to provide proven clinical benefit
* ECOG Performance Status 0 to 2
* Adequate organ function as defined by pre-specified laboratory values
* Life expectancy > 3 months
* Women of child-bearing potential (or males with female partners of child-bearing potential) must agree to use adequate contraceptive measures throughout the study and for 90 days following last dose

Key Exclusion Criteria:

* Has not completed appropriate wash-out timeframes of prior anti-cancer treatments
* Has ongoing toxicities from prior anti-cancer treatments
* Has symptomatic or uncontrolled neurologic disease
* Has active and clinically significant bacterial, fungal or viral infection
* Cannot avoid use of moderate or strong CYP3A4 inhibitors or inducers; CYP2C19 substrates or OAT2 substrates with narrow therapeutic index; or drugs that prolong the QT interval throughout the study
* Has previously received a total anthracycline dose ≥ 360mg/m2 doxorubicin or equivalent
* Has a history of serious cardiac conditions or pulmonary or cerebrovascular events within 6 months of first dose
* Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of dose limiting toxicities | 28 days
  Frequency and type of dose limiting toxicities associated with each dose level of BTM-3566
Frequency and severity of adverse events | Through study completion, estimated 2 years
  Frequency and severity of adverse events according to NCI-CTCAE v 5.0

SECONDARY OUTCOMES:
Pharmacokinetic properties of BTM-3566 | 30 days
  Plasma concentration of BTM-3566 at each time point
Clinical activity of BTM-3566 | Through study completion, estimated 2 years
  Objective Response Rate by RECIST 1.1
Clinical activity of BTM-3566 | Through study completion, estimated 2 years
  Progression Free Survival per RECIST 1.1 principles
Clinical activity of BTM-3566 | Through study completion, estimated 2 years
  Overall Survival
Clinical activity of BTM-3566 | Through study completion, estimated 2 years
  Clinical Benefit Rate (proportion of patients having at least stable disease) according to RECIST 1.1 principles
Clinical activity of BTM-3566 | Through study completion, estimated 2 years
  Duration of Response, per RECIST 1.1 principles

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NEXT Houston, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
This is an exploratory proof of concept study with no formal hypothesis testing and may not be suitable for publication in a peer-reviewed journal.